CLINICAL TRIAL: NCT04783441
Title: Continuous Glucose Monitoring (CGM) to Improve Glycemic Control in Kidney Transplant Recipients
Brief Title: Use of CGM in Kidney Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1554226
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant; Complications; Diabetes Mellitus, Type 2; Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: We propose a single-center, prospective, randomized study comprising 2 study arms. They will be randomized in a stratified fashion. Stratification will be according to whether or not they are on prednisone and their estimated glomerular filtration rate. This is to ensure that both arms are populated by equal numbers of patients with prednisone and with worse renal function
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous glucose monitoring (CGM) (Active Comparator): Those in the intervention arm will wear a continuous glucose monitoring device. They only need to perform blood glucose fingersticks if the CGM transmission is lost for a prolonged period of time or in cases of hypo- or hyperglycemia when symptoms don't align with blood glucose readings.
  Interventions: Device: Dexcom G6
- Self monitoring of blood glucose (fingersticks) (Placebo Comparator): The control arm will remain on standard-of-care SMBG while the intervention arm will use their CGM. The control arm utilizing SMBG will be required to have at minimum 4 glucose checks per day.
  Interventions: Device: Dexcom G6 blinded sensor

INTERVENTIONS:
Device: Dexcom G6 — access to continuous glucose monitoring in the Dexcom G6 arm 24/7
  Arms: Continuous glucose monitoring (CGM)
Device: Dexcom G6 blinded sensor — retrospective access to continuous glucose profile after 10 days of wear
  Arms: Self monitoring of blood glucose (fingersticks)

SUMMARY:
The investigators want to study the impact CGM (continuous glucose monitoring) has on patients glycemic control as determined by time in range (TIR 70-180 mg/dL) in the Diabetic Kidney Transplant population.

DETAILED DESCRIPTION:
Diabetes is one of the leading causes of End Stage Renal Disease (ESRD). Kidney transplantation is the best form of renal replacement therapy to date but requires that recipients of transplant organs maintain a complicated medication regimen in order to prevent graft loss. Their medications include lifelong immunosuppression, anti-microbials and other maintenance medications (i.e., anti-hypertensives, heart-protective regimens, bowel care, vitamins and pain medications).

For many transplant patients, glycemic control in the immediate post-operative period can be an additional challenge. Glycemic control may be hindered by recent surgery, corticosteroids, immunosuppressants, altered nutritional intake and reduced mobility.

Diabetes professional organizations such as the American Diabetes Association (ADA) and the American Association of Clinical Endocrinologists (AACE) recommend continuous glucose monitoring (CGM) for anyone on intensive insulin therapy. The biggest benefit of CGM is not just the actual glucose value, but also its direction and rate of change. CGM data can also be downloaded and reflect patterns of glycemic control throughout the day and night, including not only the average blood glucose but also time-in-range (TIR) and degrees of glycemic variability. This can help identify unnotified nightly hypoglycemia or hyperglycemia and help titrate medications to achieve better glycemic control. Self-Management of blood glucose (SMBG) is a key component in effective glycemic management, but it places a large burden on the patient. Prior to CGM, SMBG was the only option to measure daily blood glucose fluctuations, but it is an imperfect tool. For patients on insulin, a blood glucose is checked at minimum 4 times per day, prior to meals and at bedtime. Additionally, the utility of SMBG can be endangered by patient decision making, the ability to check blood glucose, adherence to testing regimen, error due to poor testing technique, inadequate blood supply, contamination on fingers, or inaccuracy of some systems.

Numerous studies have shown the clinical benefit of CGM in the type-1 diabetes (T1D) and type-2 diabetes (T2D) populations (ref: Beck, Olafsdottir). The DIAMOND group (Beck) showed that CGM improved HBA1C and reduced hyperglycemia (BG>180). Patients wearing the CGM had high satisfaction scores and low perceived burden. CGM is still a new tool outside of the Type 1 Diabetes population but may have significant benefits for any patient on insulin. In Feb 2019 an international guideline on TIR (defined as blood glucose of 70-180 mg/dL) was published and TIR may become a new standard for assessing glycemic control.

The investigators research focuses on TIR and the benefits of CGM in the kidney transplant population. This can be essential for timely adjustments of insulin dosages when dealing with glycemic derangements and steroid induced hyperglycemia. CGM can provide an immense opportunity for a continuous 24/7 view of glucose values, glycemic variability, direction of change and unrecognized blood glucose levels during nighttime, and influence of food and activity on blood glucose values. In addition to the metrics described; the glucose management indicator (GMI) or also named estimated A1C (eA1C) is a measure converting the mean glucose from CGM using a formula derived from glucose readings from a population of individuals, into an estimate of a simultaneously measured laboratory A1C, this value may serve as an additional tool in assessing glycemic control. In conclusion: the use of a CGM can aid the provider and care team in better titration of insulin and medication regimen adjustment. This research hopes to give insight in a very complex population that has not had access to CGM before.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. Received a kidney transplant within the past year with functioning kidney (eGFR > 30 mL/min
3. Person with Type 2 Diabetes and on insulin
4. Access to home wi-fi connection

Exclusion Criteria:

1. Person with Type 1 Diabetes
2. Patients taking hydroxyurea
3. Patient unable to wear the Dexcom G6 device at all times for any reason
4. Must be able to test blood glucose with meter 4x a day when on blinded CGM.
5. Presence of clinically significant visual or cognitive impairment
6. Illiterate
7. Prisoners
8. Women who are pregnant, who plan to become pregnant during the course of the study, or who are breastfeeding
9. Presence of clinically unstable cardiovascular disease
10. Active malignancy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in Range (70-180 mg/dl) | 70 days
  1) Time in Range: Number of minutes per day or percentage of time that glucose levels are in low (BG<70), target (BG 70-180), high (BG >180) or very high (BG>250) ranges.

SECONDARY OUTCOMES:
Glycemic variability | 70 days
  assessed by the Coefficient of Variation (Glucose standard deviation divided by mean glucose). % CV is a standardized measure that assesses the magnitude of glucose variability
CGM satisfaction questionnaire (10 questions) | up to 70 days
  score on CGM questionnaire (1 = lowest and 5 = highest)
Adherence to Diabetic Diet | up to 70 days
  Use of ASA24 online 24 hr dietary recall at 3 times throughout the study
Incidence of all-cause emergency room utilization and rehospitalizations | 70 days
  during the study period (70 days)
Incidence of post-transplant infections during study period | 70 days
  during the study period (70 days)

OTHER OUTCOMES:
safety endpoint Hypoglycemia | 70 days
  Hypoglycemia risk will be assessed as percentage of time below range (BG<70 mg/dl) and very low (BG <54 mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Ling Chen, MD, Study Director — UCDavis Transplant Nephrology
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck RW, Riddlesworth TD, Ruedy K, Ahmann A, Haller S, Kruger D, McGill JB, Polonsky W, Price D, Aronoff S, Aronson R, Toschi E, Kollman C, Bergenstal R; DIAMOND Study Group. Continuous Glucose Monitoring Versus Usual Care in Patients With Type 2 Diabetes Receiving Multiple Daily Insulin Injections: A Randomized Trial. Ann Intern Med. 2017 Sep 19;167(6):365-374. doi: 10.7326/M16-2855. Epub 2017 Aug 22. PMID 28828487
- [Background] Beck RW, Riddlesworth T, Ruedy K, Ahmann A, Bergenstal R, Haller S, Kollman C, Kruger D, McGill JB, Polonsky W, Toschi E, Wolpert H, Price D; DIAMOND Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Adults With Type 1 Diabetes Using Insulin Injections: The DIAMOND Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):371-378. doi: 10.1001/jama.2016.19975. PMID 28118453
- [Background] Olafsdottir AF, Polonsky W, Bolinder J, Hirsch IB, Dahlqvist S, Wedel H, Nystrom T, Wijkman M, Schwarcz E, Hellman J, Heise T, Lind M. A Randomized Clinical Trial of the Effect of Continuous Glucose Monitoring on Nocturnal Hypoglycemia, Daytime Hypoglycemia, Glycemic Variability, and Hypoglycemia Confidence in Persons with Type 1 Diabetes Treated with Multiple Daily Insulin Injections (GOLD-3). Diabetes Technol Ther. 2018 Apr;20(4):274-284. doi: 10.1089/dia.2017.0363. Epub 2018 Apr 2. PMID 29608107
- [Background] Edelman SV, Argento NB, Pettus J, Hirsch IB. Clinical Implications of Real-time and Intermittently Scanned Continuous Glucose Monitoring. Diabetes Care. 2018 Nov;41(11):2265-2274. doi: 10.2337/dc18-1150. PMID 30348844
- [Background] Saisho Y. Use of Diabetes Treatment Satisfaction Questionnaire in Diabetes Care: Importance of Patient-Reported Outcomes. Int J Environ Res Public Health. 2018 May 9;15(5):947. doi: 10.3390/ijerph15050947. PMID 29747423
- [Background] Garber AJ, Handelsman Y, Grunberger G, Einhorn D, Abrahamson MJ, Barzilay JI, Blonde L, Bush MA, DeFronzo RA, Garber JR, Garvey WT, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Perreault L, Rosenblit PD, Samson S, Umpierrez GE. CONSENSUS STATEMENT BY THE AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY ON THE COMPREHENSIVE TYPE 2 DIABETES MANAGEMENT ALGORITHM - 2020 EXECUTIVE SUMMARY. Endocr Pract. 2020 Jan;26(1):107-139. doi: 10.4158/CS-2019-0472. No abstract available. PMID 32022600
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S98-S110. doi: 10.2337/dc20-S009. PMID 31862752
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Longo R, Sperling S. Personal Versus Professional Continuous Glucose Monitoring: When to Use Which on Whom. Diabetes Spectr. 2019 Aug;32(3):183-193. doi: 10.2337/ds18-0093. PMID 31462872
- [Background] American Diabetes Association. 7. Diabetes Technology: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S77-S88. doi: 10.2337/dc20-S007. PMID 31862750